CLINICAL TRIAL: NCT01139125
Title: An Open Trial of Cysteamine Treatment in Schizophrenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped after 4 years of recruitment difficulties.
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Dr. Peter F. Buckley, Dean of the Medical College at Georgia Health Sciences University, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAC09-04-276
Record Dates: First submitted 2010-05-12; First posted 2010-06-08 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Schizophrenia; Schizoaffective
MeSH Terms: conditions — Schizophrenia | interventions — Cysteamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cystagon, Cysteamine Bitartrate (Experimental): We are examining the safety and efficacy of this medication on the treatment of schizophrenia patients.
  Interventions: Drug: (Cystagon) Cysteamine Bitartrate

INTERVENTIONS:
Drug: (Cystagon) Cysteamine Bitartrate — Cysteamine Bitartrate 300mg/day to 2100mg/day over a 4 month period. Number of cycles: until progression or unacceptable toxicity develops.

SUMMARY:
The purpose of this study is to determine the tolerability of the medication cysteamine bitartrate on schizophrenia patients and to evaluate the effect of the medication on the symptoms of schizophrenia.

DETAILED DESCRIPTION:
Despite the availability of numerous antipsychotics, the treatment of schizophrenia is very unsatisfactory. Many patients have persistent positive psychotic symptoms or negative symptoms despite treatment, and any improvement in cognitive function is small. New approaches to the pharmacotherapy of schizophrenia that are not based primarily on dopaminergic blockade are needed.

The rationale for a trial of cysteamine comes from the evidence that cysteamine increases brain concentrations of brain-derived neurotrophic factor.

We will conduct an open-label study of tolerability and efficacy of cysteamine as an adjunct to second-generation antipsychotics in schizophrenia and schizoaffective subjects with partially responsive symptoms.

Our objectives are to determine the safety and tolerability of cysteamine administered as an adjunct to second-generation antipsychotic drugs in adult outpatients with partially-responsive schizophrenia. Additionally, we are evaluating the effect of cysteamine on the positive and negative symptoms of schizophrenia as measured by changes in the Positive and Negative Symptom Scale (PANSS), and on cognitive impairment as measured by the Brief Assessment of Cognition in Schizophrenia (BACS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* 18-60 years of age
* Residual symptoms, as defined by both 1 & 2:

  1. At least one PANSS positive symptom item score > 4, or at least two items with a score > 3
  2. At least one PANSS negative symptom item score > 4, or at two items with a score > 3
* No clinically significant change in symptoms for at least one month
* On the same psychotropic medication(s) > 2 weeks
* Taking a second-generation antipsychotic (olanzapine, risperidone, quetiapine, ziprasidone, aripiprazole, or clozapine)
* Provision of written informed consent

Exclusion Criteria:

* Meets criteria for current major depressive disorder
* Abnormal hepatic function (AST or ALT > 2.5 X the upper limit of normal, or bilirubin > 1.5 X the upper limit of normal)
* Abnormal renal function (BUN or creatinine > 1.5 X the upper limit of normal)
* Presence of any unstable or untreated medical disorder
* Any history of seizure disorder, HIV, or diagnosis of AIDS
* Any abnormal lab test result that is judged to be clinically significant by the investigators
* Pregnancy, breast feeding, or female and of child-bearing potential who is not using any contraceptive method
* Present danger to self or others

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Buckley, M.D., Principal Investigator — Augusta University
Locations (2):
- United States (2):
  - Georgia Health Sciences University - Dept of Psychiatry, Augusta, Georgia
  - Georgia Regents University- Dept of Psychiatry, Augusta, Georgia

RESULTS

PARTICIPANT FLOW:
Groups:
- Cystagon (Cysteamine Bitartrate): Subjects were expected to take cystagon (cysteamine bitarate)14 capsules per day (4 at 7:00 am, 3 at 12:00 pm, 4 at 5:00 pm and 3 at 10:00pm) for 16 weeks.
Period: Overall Study
Arm/Group | Cystagon (Cysteamine Bitartrate)
Started | 3
Completed | 2
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Cystagon: One black male and two white males started the study
Arm/Group | Cystagon
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety and Efficacy
Description: We are measuring if this medication is appropriate for use in schizophrenia patients.
Time Frame: 4 months
Groups:
- Cystagon: Subjects are required to take 14 capsules per day for 16 weeks
Arm/Group | Cystagon
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Cystagon: Subjects taking 14 capsules per day for 16 weeks
Arm/Group | Cystagon
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cystagon (N=3)
Jaw Hair Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Recruitment challenges for this study are the number of pills that the subjects are required to take during treatment and the reported foul body odor that the subjects complianed of and was also noted by the Investigator and research staff.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No